CLINICAL TRIAL: NCT00596921
Title: Bedside Ultrasound Measurement of the Inferior Vena Cava Correlates to Central Venous Pressure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: COL Robert De Lorenzo, Brooke Army Medical Center
Other Study IDs: C.2008.029; CIRO.2008111
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2008-01

CONDITIONS: Shock; Hypovolemia; Hypervolemia
Keywords: Ultrasonography; Central Venous Pressure; Noninvasive monitoring; Shock; Resuscitation
MeSH Terms: conditions — Shock; Hypovolemia; Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study proposes to examine the correlation of central venous pressure to measures of the diameter of the inferior vena cava as determined by bedside ultrasonography.

DETAILED DESCRIPTION:
Central venous pressure (CVP) is a key physiologic estimate of preload, which in turn helps define the vascular fluid status. It is a particularly important parameter to measure in critically ill and injured patients who may require resuscitation. Unfortunately, measurement of the CVP requires invasive central venous catheters which can be difficult or time-consuming to insert. A non-invasive means of inferring the CVP would provide clinicians with an alternative. Preliminary data suggests that the diameter of the vena cava may reflect the CVP. Ultrasonography can provide reliable measures of internal body structures including the vena cava, and therefore may be useful in this regard. Collecting simultaneous values of vena cava diameter and CVPs will allow for the identification and quantification of correlation.

ELIGIBILITY:
Inclusion Criteria:

* CVP or right heart catheter that is already in place and functioning properly

Exclusion Criteria:

* Supine position or placement of ultrasound probe on abdomen is contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with central venous monitoring in place.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)

PRIMARY OUTCOMES:
Bedside ultrasound measurement of the diameter of the inferior vena cava and simultaneously measured central venous pressure. | Cross-sectional

SECONDARY OUTCOMES:
Anatomic view and phase of respiration at the time of measurements. | Cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Robert A De Lorenzo, MD, Principal Investigator — Brooke Army Medical Center